CLINICAL TRIAL: NCT01789723
Title: An Open Label, Multicenter, Dose Finding, Phase 1 Study of Fusilev® (Levoleucovorin) to Prevent or Reduce Mucositis in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma Receiving Folotyn® (Pralatrexate)
Brief Title: Phase 1 Study of Fusilev to Prevent or Reduce Mucositis in Patients With Non-Hodgkin's Lymphoma Receiving Folotyn
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPI-FUS-12-102
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Levoleucovorin; 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Fusilev - 10 doses (Experimental): Fusilev: 5 mg/m2 QID, starting on Day 2 (24 ± 3 hours after Folotyn dose) for a total of 10 doses Day 2: 4 doses Day 3: 4 doses Day 4: 2 doses.
  Folotyn: 30 mg/m2 once weekly for 6 weeks
  Interventions: Drug: Fusilev; Drug: Folotyn
- Cohort 2: Fusilev - 6 doses (Experimental): Fusilev: 5 mg/m2 BID, on Days 2 (24 ± 3 hours after Folotyn dose), 3, and 4.
  Folotyn: 30 mg/m2 once weekly for 6 weeks
  Interventions: Drug: Fusilev; Drug: Folotyn
- Cohort 3: Fusilev - 4 doses (Experimental): 5 mg/m2 BID, on Days 2 (24 ± 3 hours after Folotyn dose) and 3.
  Folotyn: 30 mg/m2 once weekly for 6 weeks
  Interventions: Drug: Fusilev; Drug: Folotyn
- Cohort 4: Fusilev - 2 doses (Experimental): 5 mg/m2 BID, on Day 2 (24 ± 3 hours after Folotyn dose.
  Folotyn: 30 mg/m2 once weekly for 6 weeks
  Interventions: Drug: Fusilev; Drug: Folotyn
- Cohort 5: Fusilev - 1 dose (Experimental): Fusilev: 5 mg/m2 once on Day 2.
  Folotyn: 30 mg/m2 once weekly for 6 weeks
  Interventions: Drug: Fusilev; Drug: Folotyn

INTERVENTIONS:
Drug: Fusilev — Fusilev will be administered by IV push (3-5 minutes) at a dose of 5 mg/m2. Fusilev administration, QID or BID will start 24 ± 3 hours after Folotyn administration depending on the dose cohort.
  Other Names: Fusilev - (Levoleucovorin)
Drug: Folotyn — A cycle of Folotyn treatment is 7 weeks, 6 weeks of treatment followed by 1 week of rest.
  Other Names: Folotyn - (Pralatrexate)

SUMMARY:
The purpose of this study is determine the optimal dose and schedule of Fusilev to prevent or reduce Mucositis in patients with Non-Hodgkin's Lymphoma receiving Folotyn treatment.

DETAILED DESCRIPTION:
This is an open label, uncontrolled, nonrandomized, multicenter, dose finding, Phase 1 study primarily to determine the optimal dose and schedule of Fusilev to prevent or reduce Folotyn-related Grade 3 or higher oral Mucositis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Patients with relapsed or refractory NHL who are eligible for Folotyn treatment. Patient has histologically/cytologically confirmed, measurable (lesion or node ≥ 2 cm by computed tomography [CT]
* Progressive disease or persistent disease after at least 1 prior treatment
* ECOG performance status ≤ 2
* Adequate hematological, hepatic, and renal function

Exclusion Criteria:

* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix)
* Congestive heart failure
* Uncontrolled hypertension
* Known human immunodeficiency virus (HIV)-positive diagnosis
* Active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the patient to receive protocol treatment
* Major surgery within 14 days of enrollment
* Pregnant or breast-feeding women
* Symptomatic central nervous system (CNS) metastases or lesions for which treatment is required. Patients who received prophylactic CNS treatment are eligible
* Previous exposure to pralatrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Optimal dose and schedule of Fusilev to prevent or reduce mucositis | Up to 8 weeks
  The patient will be seen in the clinic for an oral mucositis assessment at baseline. During the 6 weeks of Folotyn treatment, oral mucositis assessment will be performed weekly prior to each Folotyn dose and again on Day 4 (prior to the Fusilev dose when applicable) by a qualified health care professional. Patients will complete an Oral Mucositis Daily Questionnaire (OMQD) starting at Day 1 of Week 1 and ending at the End of Treatment Visit.

SECONDARY OUTCOMES:
Impact of Fusilev on Folotyn related Oral Mucositis | 7 weeks
  To determine the impact of Fusilev on the number of Folotyn-related dose modifications secondary to oral mucositis To determine the impact of Fusilev on the frequency of Folotyn-related oral mucositis To determine the impact of Fusilev on the number of Folotyn doses delivered
Relationship between Fusilev use and oral mucositis | 7 weeks
  To determine the relationship between Fusilev use and oral mucositis as a function of the pretreatment homocysteine (HCY) and methylmalonic acid (MMA) levels

OTHER OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  To determine overall response rate (ORR) of Folotyn in relapsed or refractory Non-Hodgkin's lymphoma other than PTCL

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Sawas, MD, Principal Investigator — Columbia University